CLINICAL TRIAL: NCT05639712
Title: Understanding Opioid Use Before and After Surgery in Norway: A Prospective Multicenter Study and Randomized Double-blind Controlled Study
Brief Title: Affective Effects of Pre-surgery Opioids: a Randomized, Doubleblind Placebo-controlled Trial
Acronym: AFFECT2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre VikenHF Kongsberg Sykehus (Other)
Responsible Party: Principal Investigator, Harald Lenz, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AFFECT2 Version 2, 04.11.2022; 2022-002938-13 (EudraCT Number)
Record Dates: First submitted 2022-11-17; First posted 2022-12-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use; Affective Symptoms
MeSH Terms: conditions — Affective Symptoms | interventions — Morphine; Oxycodone; Fentanyl

STUDY DESIGN:
Intervention Model Description: The patient will be randomized to 1 of 10 arms: Placebo (saline 0.9%), morphine 2.5 - 5 - 10 mg, oxycodone 2.5 - 5 -10 mg, or fentanyl 0.025 - 0.05 - 0.1 mg iv.
Who Masked: Participant, Investigator
Masking Description: Randomization sequences will be generated prior to the first enrolment of the amended protocol by an independent group (Clinical trails unit- OUS) not affiliated with the present study.
  The drug will be prepared after opening an opaque envelope on the day of surgery by a nurse not participating in the study. The syringe with the drug will be labeled with a code number and handed to the study nurse or doctor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Placebo (Placebo Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of placebo (0.9% NaCl intravenously). This is carried out on the operating table right before anesthesia
  Interventions: Drug: Placebo
- Morphine 2.5 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of morphine 2.5 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Morphine 2.5 mg i.v.
- Morphine 5 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of morphine 5 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Morphine 5 mg i.v.
- Morphine 10 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of morphine 10 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Morphine 10 mg i.v.
- Oxycodone 2.5 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of oxycodone 2.5 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Oxycodone 2.5 mg i.v.
- Oxycodone 5 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of oxycodone 5 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Oxycodone 5 mg i.v.
- Oxycodone 10 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of oxycodone 10 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Oxycodone 10 mg i.v.
- Fentanyl 0.025 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of fentanyl 0.025 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Fentanyl 0.025 mg i.v.
- Fentanyl 0.05 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of fentanyl 0.05 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Fentanyl 0.05 mg i.v.
- Fentanyl 0.1 mg (Active Comparator): The patient is given standardized questions about their well-being and affective state before and after the administration of fentanyl 0.1 mg intravenously. This is carried out on the operating table right before anesthesia
  Interventions: Drug: Fentanyl 0.1 mg i.v.

INTERVENTIONS:
Drug: Placebo — The patient is given standardized questions about their well-being and affective state before and after the administration of placebo intravenously. This is carried out on the operating table right before anesthesia
  Other Names: 0.9% NaCl , Natriumklorid 9 mg/ml, Hameln (ATC code: B05B B01)
  Arms: Placebo
Drug: Morphine 2.5 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of 2.5 mg morphine intravenously. This is carried out on the operating table right before anesthesia
  Other Names: Morphine, Orion (ATC code: N02A A01)
  Arms: Morphine 2.5 mg
Drug: Morphine 5 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of morphine 5 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Morphine, Orion (ATC code: N02A A01)
  Arms: Morphine 5 mg
Drug: Morphine 10 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of morphine 10 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Morphine, Orion (ATC code: N02A A01)
  Arms: Morphine 10 mg
Drug: Oxycodone 2.5 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of oxycodone 2.5 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Oxycodone, Hameln (ATC code: N02A A05)
  Arms: Oxycodone 2.5 mg
Drug: Oxycodone 5 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of oxycodone 5 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Oxycodone, Hameln (ATC code: N02A A05)
  Arms: Oxycodone 5 mg
Drug: Oxycodone 10 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of oxycodone 10 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Oxycodone, Hameln (ATC code: N02A A05)
  Arms: Oxycodone 10 mg
Drug: Fentanyl 0.025 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of fentanyl 0.025 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Fentanyl, Hameln (ATC code: N01A H01)
  Arms: Fentanyl 0.025 mg
Drug: Fentanyl 0.05 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of fentanyl 0.05 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Fentanyl, Hameln (ATC code: N01A H01)
  Arms: Fentanyl 0.05 mg
Drug: Fentanyl 0.1 mg i.v. — The patient is given standardized questions about their well-being and affective state before and after the administration of fentanyl 0.1 mg intravenously . This is carried out on the operating table right before anesthesia
  Other Names: Fentanyl, Hameln (ATC code: N01A H01)
  Arms: Fentanyl 0.1 mg

SUMMARY:
1. To investigate and compare the affective short-term effects of opioid drugs: morphine, oxycodone and fentanyl, administered to the patients before the induction of general anesthesia.
2. Charting opioid use after surgery in patients treated at hospitals in Norway
3. Identify predictors for postoperative opioid use and persistent pain

DETAILED DESCRIPTION:
The aim of the present study is to assess and compare, with a randomized, double-blind placebo-controlled trial, the affective effects of three commonly used opioid analgesics (Morphine, oxycodone and fentanyl) administered in three different doses before surgery in a clinical setting associated with physiological and psychological stress.

As a starting point, we have conducted an observational quality control study on peri-operative opioid pain management in day surgery patients.

Quality control study - a pilot study In this observational quality control study, we measured acute effects of the opioid agonist Remifentanil (effect site concentration 5ng/ml, Minto model) in day surgery patients on the operating table at Kongsberg hospital. Patients rated their levels of "feeling good" and "anxious" on a 0-10 numerical rating scale (NRS) immediately before and 1 minute after receiving remifentanil infusion. They also rated drug-specific effects such as "feeling high", "liking the drug effects" and their "level of drug-related discomfort". Moreover, we collected data on postoperative opioid use and pain during recovery through a telephone interview on the day following the surgery. The study was conducted with the usual standard hospital treatment and as such, did not interfere with the patients' medical procedures. All the procedures were approved by the data protection officer at Kongsberg Hospital, and all included patients signed informed consent on the day of surgery.

In the weeks prior to surgery participants received a questionnaire to assess their pain levels, nervousness and demographics as part of the hospital's standard procedure. On the day of surgery, approximately 30 min before surgery (T2) patients were asked to fill in questionnaires to assess mood, pain and prior opioid use. One minute before and one minute after opioid ( administration (T3), the patient was asked to rate mood, anxiety, drug liking and drug related discomfort. On the day following surgery patients were contacted by phone to assess their mood, pain and pain interference, as well as their pain relief strategies in the last 24h (e.g. use of provided analgesics).

160 patients were included in the pilot quality control study. The results of the pilot study show that patients report a clear feeling of 'drug high' after remifentanil infusion. Surprisingly, however, the opioid analgesic induced only a weak reduction of anxiety, and the majority of patients reported feeling worse or equally good, but not better, after the infusion. In the postoperative phone interview, many patients tell us they have not used any of the opioid drugs prescribed for at-home pain relief during the first 24 hours are recovering at home. Stated reasons include a fear of addiction, as well as a wish to keep the analgesics in case of breakthrough/peak pain at a later stage. These preliminary results do not support the opioid pre-induction procedure as an effective manner to produce pre-surgery stress relief. It might be possible that the subjective perception of stress relief does not match the physiological relief reaction to stress.

On the basis of these intriguing, preliminary findings, we will now conduct a more comprehensive randomized double-blind controlled study comparing different classes of pre-surgical opioid analgesics on the subjective and physiological affective reactions in an acute stress clinical situation in Norway.

Possible participants of the AFFECT2 RCT (randomized controlled trial) will also be asked if they wish to join a parallel longitudinal study conducted in collaboration with the University of Oslo (UiO) in which we will collect and analyse data on relevant pre-surgery risk factors for problematic opioid use, and to quantify opioid-induced analgesia before and after surgery using prescription registry data.

ELIGIBILITY:
Inclusion Criteria:

- Health status ASA1 (American Society of Anesthesiologists physical status) or ASA2 as categorised by a medical doctor at the hospital based on medical history, physical examination, laboratory test etc. unrelated to the current study.

ASA1 and ASA2 (ASA1 is defined as "Healthy, non-smoking, no or minimal alcohol use" and ASA2 is defined as "Mild diseases only without substantive functional limitations). Being eligible for day surgery means participants are overtly healthy as determined by clinical staff.

* The participant is considered as eligible for the use of fentanyl, morphine and oxycodone by a medical doctor at the hospital, based on an overall assessment of the psychiatric and somatic condition, used medical drugs, regarding possible interactions and contraindications for the use of the study medicaments.
* Body weight and body mass index (BMI) within the range 18-35 kg/m2 (inclusive).
* Capable of giving signed informed consent as which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Having good verbal communication skills in Norwegian.
* Patients undergoing planned day surgery with general anesthesia (outpatient sample).
* Orthopedic, rectal, gynecological, hand and foot surgery, and minor vascular procedures.
* Inpatients undergoing planned gynecological and orthopedic surgery.
* Hysterectomy, laparoscopic ovariectomy, lumbal herniotomy and other related procedures.
* Minor gastrointestinal surgery

Exclusion Criteria:

1. Known allergic reactions to morphine, oxycodone,or fentanyl. Known allergic reactions to any of the incredients described in the SPC, pt 6.1.
2. Severe chronic obstructive lung disease,
3. Cor pulmonale,
4. Severe bronchial asthma,
5. Severe respiratory failure with hypoxemia and hypercapnia
6. Moderate to severe hepatic impairment,
7. Moderate to severe kidney failure
8. Acute abdomen
9. Increased brain pressure
10. Head trauma
11. Use of MAO blockers in the last two weeks
12. Hypovolemia
13. Hypotension
14. Myasthenia gravis
15. Any other health status not corresponding to ASA1 or ASA2. This includes patients with severe disease burden, major psychiatric disorders that could interfere with the procedures and communication.
16. Pregnancy. Women of childbearing potential defined as all premenopausal female (a postmenopausal state is defined as no menses for 12 months without an alternative medical cause) will be asked if they are pregnant.
17. Breastfeeding women.
18. Illegal drugs use like opioids, cocaine and amphetamine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Anxious | 8-10 minutes
  Asking the patient of feeling anxious; Numeric rating scale 0 -10 prior opioid and post opioid intravenously (or placebo). 0=not anxious and 10=feeling extremely anxious
Relaxed | 8-10 minutes
  Asking the patient of feeling relaxed. Numeric rating scale 0 -10 prior opioid and post opioid intravenously (or placebo). 0=not relaxed and 10=very relaxed.
Pain level | 8-10 minutes
  Asking the patient of pain level. Numeric rating scale 0 -10 prior opioid and post opioid intravenously (or placebo). 0=no pain and 10= worst pain imaginable
Good | 8-10 minutes
  Asking the patient of feeling good. Numeric rating scale 0 -10 prior opioid and post opioid intravenously (or placebo). 0=feeling no good and 10= feeling very good.
Dizzy | 2-4 minutes
  Asking the patient of feeling dizzy. Numeric rating scale 0-10 post opioid intravenously (or placebo). 0=feeling not dizzy and 10=feeling very dizzy.
Sedated | 2-4 minutes
  Asking the patient of feeling sedated. Numeric rating scale 0-10 post opioid intravenously (or placebo). 0=feeling not sedated and 10=feeling very sedated.
Feeling high, Numeric rating scale 0 -10 | 2-4 minutes
  Asking the patient of feeling high. Numeric rating scale 0-10 post opioid intravenously (or placebo). 0=feeling not high and 10=feeling very high.
Euphoric | 2-4 minutes
  Asking the patient of feeling high. Numeric rating scale 0-10 post opioid intravenously (or placebo). 0=feeling not euphoric and 10=feeling very euphoric.
Drug liking | 2-4 minutes
  Asking the patient of drug liking. Numeric rating scale 0-10 post opioid intravenously (or placebo). 0=feeling not drug liking and 10=feeling very drug liking.
Drug disliking | 2-4 minutes
  Asking the patient of drug disliking. Numeric rating scale 0-10 post opioid intravenously (or placebo). 0=feeling not drug disliking and 10=feeling very drug disliking.

OTHER OUTCOMES:
Heart rate | 10 min
  beats/min prior opioid and post opioid intravenously
Heart rate variability | 10 min
  Heart rate variability (HRV) prior opioid and post opioid intravenously

CONTACTS AND LOCATIONS:
Overall Officials: Gernot Ernst, MD,PhD, Principal Investigator — Kongsberg Hospital, Vestre Viken Health Trust Norway
Locations (1):
- Harald Lenz, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angst MS, Lazzeroni LC, Phillips NG, Drover DR, Tingle M, Ray A, Swan GE, Clark JD. Aversive and reinforcing opioid effects: a pharmacogenomic twin study. Anesthesiology. 2012 Jul;117(1):22-37. doi: 10.1097/ALN.0b013e31825a2a4e. PMID 22713632
- [Background] Astuto, M., & Lauretta, D. (2009). Anesthesia Induction. In M. Astuto (Ed.), Basics (pp. 85-99). Milano: Springer Milan.
- [Background] Bershad AK, Miller MA, Norman GJ, de Wit H. Effects of opioid- and non-opioid analgesics on responses to psychosocial stress in humans. Horm Behav. 2018 Jun;102:41-47. doi: 10.1016/j.yhbeh.2018.04.009. Epub 2018 Apr 24. PMID 29673620
- [Background] Bjerkeset O, Romild U, Smith GD, Hveem K. The associations of high levels of C-reactive protein with depression and myocardial infarction in 9258 women and men from the HUNT population study. Psychol Med. 2011 Feb;41(2):345-52. doi: 10.1017/S0033291710000887. Epub 2010 May 6. PMID 20444310
- [Background] Choudhary P, Dutta A, Sethi N, Sood J, Rai D, Gupta M. Pre-induction fentanyl dose-finding study for controlled hypotension during functional endoscopic sinus surgery. Indian J Anaesth. 2019 Aug;63(8):653-659. doi: 10.4103/ija.IJA_866_18. PMID 31462812
- [Background] Colasanti A, Rabiner EA, Lingford-Hughes A, Nutt DJ. Opioids and anxiety. J Psychopharmacol. 2011 Nov;25(11):1415-33. doi: 10.1177/0269881110367726. Epub 2010 Jun 8. PMID 20530588
- [Background] Courtwright, D. T. (2001). Dark Paradise: A History of Opiate Addiction in America. Cambridge MA: Harvard University Press.
- [Background] Dale O, Moksnes K, Kaasa S. European Palliative Care Research Collaborative pain guidelines: opioid switching to improve analgesia or reduce side effects. A systematic review. Palliat Med. 2011 Jul;25(5):494-503. doi: 10.1177/0269216310384902. PMID 21708856
- [Background] Deighton S, Neville A, Pusch D, Dobson K. Biomarkers of adverse childhood experiences: A scoping review. Psychiatry Res. 2018 Nov;269:719-732. doi: 10.1016/j.psychres.2018.08.097. Epub 2018 Aug 25. PMID 30273897
- [Background] Doleman B, Leonardi-Bee J, Heinink TP, Bhattacharjee D, Lund JN, Williams JP. Pre-emptive and preventive opioids for postoperative pain in adults undergoing all types of surgery. Cochrane Database Syst Rev. 2018 Dec 3;12(12):CD012624. doi: 10.1002/14651858.CD012624.pub2. PMID 30521692
- [Background] Drewes AM, Jensen RD, Nielsen LM, Droney J, Christrup LL, Arendt-Nielsen L, Riley J, Dahan A. Differences between opioids: pharmacological, experimental, clinical and economical perspectives. Br J Clin Pharmacol. 2013 Jan;75(1):60-78. doi: 10.1111/j.1365-2125.2012.04317.x. PMID 22554450
- [Background] Dutta A, Sethi N, Choudhary P, Sood J, Panday BC, Chugh PT. The impact of preinduction fentanyl dosing strategy on postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy. J Opioid Manag. 2018 Jul/Aug;14(4):283-293. doi: 10.5055/jom.2018.0460. PMID 30234925
- [Background] Evans SM, Foltin RW, Levin FR, Fischman MW. Behavioral and subjective effects of DN-2327 (pazinaclone) and alprazolam in normal volunteers. Behav Pharmacol. 1995 Mar;6(2):176-186. PMID 11224325
- [Background] Garland EL, Froeliger B, Zeidan F, Partin K, Howard MO. The downward spiral of chronic pain, prescription opioid misuse, and addiction: cognitive, affective, and neuropsychopharmacologic pathways. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2597-607. doi: 10.1016/j.neubiorev.2013.08.006. Epub 2013 Aug 26. PMID 23988582
- [Background] Helsedirektoratet. (2018). Utvikling og variasjon i kirurgisk behandling 2013-2017. Retrieved from Oslo:
- [Background] Levy N, Mills P. Controlled-release opioids cause harm and should be avoided in management of postoperative pain in opioid naive patients. Br J Anaesth. 2019 Jun;122(6):e86-e90. doi: 10.1016/j.bja.2018.09.005. Epub 2018 Oct 19. No abstract available. PMID 30915981
- [Background] Li PH, Ue KL, Wagner A, Rutkowski R, Rutkowski K. Opioid Hypersensitivity: Predictors of Allergy and Role of Drug Provocation Testing. J Allergy Clin Immunol Pract. 2017 Nov-Dec;5(6):1601-1606. doi: 10.1016/j.jaip.2017.03.035. Epub 2017 May 24. PMID 28550985
- [Background] Martel MO, Dolman AJ, Edwards RR, Jamison RN, Wasan AD. The association between negative affect and prescription opioid misuse in patients with chronic pain: the mediating role of opioid craving. J Pain. 2014 Jan;15(1):90-100. doi: 10.1016/j.jpain.2013.09.014. Epub 2013 Oct 12. PMID 24295876
- [Background] McHugh RK, Weiss RD, Cornelius M, Martel MO, Jamison RN, Edwards RR. Distress Intolerance and Prescription Opioid Misuse Among Patients With Chronic Pain. J Pain. 2016 Jul;17(7):806-14. doi: 10.1016/j.jpain.2016.03.004. Epub 2016 Apr 4. PMID 27058161
- [Background] Morean ME, de Wit H, King AC, Sofuoglu M, Rueger SY, O'Malley SS. The drug effects questionnaire: psychometric support across three drug types. Psychopharmacology (Berl). 2013 May;227(1):177-92. doi: 10.1007/s00213-012-2954-z. Epub 2012 Dec 28. PMID 23271193
- [Background] Natusch D. Equianalgesic doses of opioids - their use in clinical practice. Br J Pain. 2012 Feb;6(1):43-6. doi: 10.1177/2049463712437628. No abstract available. PMID 26516465
- [Background] Naude PJW, Roest AM, Stein DJ, de Jonge P, Doornbos B. Anxiety disorders and CRP in a population cohort study with 54,326 participants: The LifeLines study. World J Biol Psychiatry. 2018 Sep;19(6):461-470. doi: 10.1080/15622975.2018.1433325. Epub 2018 Feb 22. PMID 29376460
- [Background] Schaffer CB, Nordahl TE, Schaffer LC, Howe J. Mood-elevating effects of opioid analgesics in patients with bipolar disorder. J Neuropsychiatry Clin Neurosci. 2007 Fall;19(4):449-52. doi: 10.1176/jnp.2007.19.4.449. PMID 18070849
- [Background] Sgoifo A, Carnevali L, Alfonso Mde L, Amore M. Autonomic dysfunction and heart rate variability in depression. Stress. 2015;18(3):343-52. doi: 10.3109/10253890.2015.1045868. Epub 2015 May 25. PMID 26004818
- [Background] Sneader, W. (2005). Drug discovery : a history. Chichester: Wiley.
- [Background] Stanley TH. The history and development of the fentanyl series. J Pain Symptom Manage. 1992 Apr;7(3 Suppl):S3-7. doi: 10.1016/0885-3924(92)90047-l. PMID 1517629
- [Background] Stone AL, Becker LG, Huber AM, Catalano RF. Review of risk and protective factors of substance use and problem use in emerging adulthood. Addict Behav. 2012 Jul;37(7):747-75. doi: 10.1016/j.addbeh.2012.02.014. Epub 2012 Feb 24. PMID 22445418
- [Background] Thomas EA, Garland EL. Mindfulness is Associated With Increased Hedonic Capacity Among Chronic Pain Patients Receiving Extended Opioid Pharmacotherapy. Clin J Pain. 2017 Feb;33(2):166-173. doi: 10.1097/AJP.0000000000000379. PMID 28060783
- [Background] Tracey I, Woolf CJ, Andrews NA. Composite Pain Biomarker Signatures for Objective Assessment and Effective Treatment. Neuron. 2019 Mar 6;101(5):783-800. doi: 10.1016/j.neuron.2019.02.019. PMID 30844399
- [Background] Wang LP, Hermann C, Westrin P. Thiopentone requirements in adults after varying pre-induction doses of fentanyl. Anaesthesia. 1996 Sep;51(9):831-5. doi: 10.1111/j.1365-2044.1996.tb12611.x. PMID 8882244

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT05639712/Prot_SAP_000.pdf